CLINICAL TRIAL: NCT04251871
Title: Effects of Traditional Chinese Medicines (TCMs) on Patients With COVID-19 Infection: A Perspective, Open-labeled, Randomized, Controlled Trial
Brief Title: Treatment and Prevention of Traditional Chinese Medicines (TCMs) on COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiaohe Xiao, Principal Investigator, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020001D
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Pneumonia Caused by Human Coronavirus (Disorder)
MeSH Terms: interventions — Oxygen; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional medicines and TCMs granules (Experimental): Conventional medicines: oxygen therapy, antiviral therapy (alfa interferon via aerosol inhalation, and lopinavir/ritonavir, 400mg/100mg, p.o, bid) for 14 days.
  Traditional Chinese Medicines (TCMs) granules: one bag, p.o, bid, for 14 days.
  Interventions: Drug: Conventional medicines (Oxygen therapy, alfa interferon via aerosol inhalation, and lopinavir/ritonavir) and Traditional Chinese Medicines (TCMs) granules
- Conventional medicines (Active Comparator): Conventional medicines: oxygen therapy, antiviral therapy (alfa interferon via aerosol inhalation, and lopinavir/ritonavir, 400mg/100mg, p.o, bid) for 14 days.
  Interventions: Drug: Conventional medicines (Oxygen therapy, alfa interferon via aerosol inhalation, and lopinavir/ritonavir)

INTERVENTIONS:
Drug: Conventional medicines (Oxygen therapy, alfa interferon via aerosol inhalation, and lopinavir/ritonavir) and Traditional Chinese Medicines (TCMs) granules — Conventional medicines: oxygen therapy, antiviral therapy (alfa interferon via aerosol inhalation, and lopinavir/ritonavir, 400mg/100mg, p.o, bid) for 14 days.
  Traditional Chinese Medicines (TCMs) granules: 20g, p.o, bid, for 14 days.
  Arms: Conventional medicines and TCMs granules
Drug: Conventional medicines (Oxygen therapy, alfa interferon via aerosol inhalation, and lopinavir/ritonavir) — Conventional medicines: oxygen therapy, antiviral therapy (alfa interferon via aerosol inhalation, and lopinavir/ritonavir, 400mg/100mg, p.o, bid) for 14 days.
  Arms: Conventional medicines

SUMMARY:
The aim of this study is to test whether Traditional Chinese Medicines (TCMs) are effective and safe for treating COVID-19 infection. After the enrolment of approximately 30 subjects, the recruitment will be paused, and planned interim analysis will be performed to preliminarily investigate the efficacy and safety of TCMs in patients infected with COVID-19.

DETAILED DESCRIPTION:
In December 2019, a cluster of patients with pneumonia in Wuhan, China, was caused by a novel betacoronavirus, which named the 2019 novel coronavirus (COVID-19). It was frequently reported that COVID-19 could be a public health crisis with high infectiousness, and it naturally spread across the country. Most of patients with COVID-19 infection were found to have non-specific symptoms including fever, cough, myalgia and fatigue. In addition, some patients were more likely to develop severe respiratory illness similar to severe acute respiratory syndrome (SARS), or even die. However, there was no timely and effective treatment of patients with COVID-19 infection. Traditional Chinese medicines (TCMs), are derived from plants and usually incorporate one or more herbs as the basic drug(s) to treat the disease. An RCT was performed to investigate TCM was effective and safe for treating COVID-19 infection. Eligible subjects will be randomized in a 1:1 ratio, and 1 subject on conventional medicines and TCMs granules for every 1 subject on conventional medicines. According to recommendations for prevention and control of pneumonia cause by COVID-19 infection from China National Health Commission, conventional medicines involve oxygen therapy and antiviral therapy (alfa interferon via aerosol inhalation, and lopinavir/ritonavir, p.o). Additionally, planned interim analysis will be performed, because the prevention and control of COVID-19 infection might affect estimated enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection case in term of laboratory evidence;
* 80 years ≥ age ≥ 14years;
* Within 72 hours after the onset of abnormalities shown by Chest radiology or several symptoms (fever and cough).

Exclusion Criteria:

* Age < 14 years or > 80 years;
* Pregnant or lactating female;
* One of the following items occurred at the enrollment: (i) respiratory failure necessitating mechanical ventilation; (ii) liver failure: total bilirubin ≥ 10mg/dL and/or severe coagulation disorders; (iii) renal function failure: although adequate circulating blood and cardiac output, urine ≤ 0.5ml/kg·h, Cr or BUN ≥ 1.5 times normal elevation;
* Intake of Chinese medicinal herbs during the past 2 weeks;
* Refused to sign an informed consent form prior to study participation;
* Unwilling and unable to comply with protocol request.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
The incidents of acute respiratory distress syndrome (ARDS) development | 14 days
  The incidence rate of acute respiratory distress syndrome (ARDS) development

SECONDARY OUTCOMES:
The time to fever resolution rate | 14 days
  Time to complete remission of fever in eligible subjects
Time to recovery of lung injury | 14 days
  improvement of chest radiographic evidence indirectly reflects recovery in patients infected with COVID-19.

OTHER OUTCOMES:
Rate of subjects who die | 28 days
  The rate of subject who die will be described.
Rate of subjects receiving systematic corticosteroids | 28 days
  The rate of subjects with severe 2019-nCoV infection who receive systematic corticosteroids will be described.
The length of hospital stays | 28 days
  The length of hospital stays
The duration of respiratory support | 28 days
  The duration of respiratory support including invasive and non-invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-he Xiao, PD., Study Director — 302 Military Hospital
Locations (1):
- The Fifth Medical Center, General Hospital of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] World Health Organization. Clinical management of severe acute respiratory infection when novel coronavirus (nCoV) infection is suspected: interim guidance. Published January 28, 2020. Accessed January 31, 2020. https://www. who.int/publications-detail/clinical-managementof- severe-acute-respiratory-infection-when-novelcoronavirus-( ncov)-infection-is-suspected
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583
- [Derived] Wang JB, Wang ZX, Jing J, Zhao P, Dong JH, Zhou YF, Yang G, Niu M, Zhao X, Jiang TJ, Bi JF, Xu Z, Zhang P, Wu D, Bai ZF, Guo YM, Yu SM, Sun YQ, Zhang ZT, Zhan XY, Li PY, Ding JB, Zhao PF, Song XA, Tang JY, He DC, Chen Z, Qin EQ, Wang RL, Xiao XH. Exploring an Integrative Therapy for Treating COVID-19: A Randomized Controlled Trial. Chin J Integr Med. 2020 Sep;26(9):648-655. doi: 10.1007/s11655-020-3426-7. Epub 2020 Jul 16. PMID 32676976